CLINICAL TRIAL: NCT01267201
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 3-Treatment, Crossover Bioavailability Study Comparing Constituted Methylprednisolone Powder For Oral Suspension 4 Mg/Ml to Methylprednisolone 32 Mg Tablet Under Fasted Conditions
Brief Title: A Study Comparing Drug Availability Of Methylprednisolone In Liquid Form Versus Methylprednisolone In Tablet Form
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0121005
Record Dates: First submitted 2010-12-13; First posted 2010-12-28 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-05

CONDITIONS: Biological Availability
Keywords: Single dose bioavailability study of methylprednisolone powder for oral suspension (4mg/mL) versus methylprednisolone tablet (32 mg)
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- POS formulation #1 (Experimental)
  Interventions: Drug: methylprednisolone
- POS formulation #2 (Experimental)
  Interventions: Drug: methylprednisolone
- commercial tablet (Active Comparator)
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — powder for oral suspension 4 mg/mL single dose (8 mL)
  Arms: POS formulation #1
Drug: methylprednisolone — powder for oral suspension 4 mg/mL singe dose (8 ml)
  Arms: POS formulation #2
Drug: methylprednisolone — tablet 32 mg single dose
  Arms: commercial tablet

SUMMARY:
A new formulation of methylprednisolone is being developed. A study is needed to determine the drug availability using the new formulation, a powder for reconstitution into a suspension, versus the current commercially available tablet formulation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2;
* a total body weight >45 kg (99 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease;
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0121005&StudyName=A%20Study%20Comparing%20Drug%20Availability%20Of%20Methylprednisolone%20In%20Liquid%20Form%20Versus%20Methylprednisolone%20In%20Tablet%20Form

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2: Single oral dose of methylprednisolone 32 milligram (mg) tablet on Day 1 in first intervention period; followed by single dose of formulation 1: methylprednisolone oral suspension 4 milligram/milliliter (mg/mL) at 32 mg (Micronized active pharmaceutical ingredient [API]) on Day 1 in second intervention period; and single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
- Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1: Single oral dose of methylprednisolone 32 mg tablet on Day 1 in first intervention period; followed by single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in second intervention period; and single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
- Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2: Single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 in first intervention period; followed by single oral dose of methylprednisolone 32 mg tablet on Day 1 in second intervention period; and single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
- Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet: Single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 in first intervention period; followed by single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in second intervention period; and single oral dose of methylprednisolone 32 mg tablet on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
- Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1: Single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in first intervention period; followed by single oral dose of methylprednisolone 32 mg tablet on Day 1 in second intervention period; and single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
- Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet: Single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 in first intervention period; followed by single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 in second intervention period; and single oral dose of methylprednisolone 32 mg tablet on Day 1 in third intervention period. A washout period of at least 2 days was maintained between each intervention period.
Period: First Intervention Period
Arm/Group | Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2 | Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1 | Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2 | Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet | Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1 | Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 2 Days)
Arm/Group | Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2 | Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1 | Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2 | Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet | Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1 | Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2 | Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1 | Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2 | Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet | Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1 | Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 2 Days)
Arm/Group | Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2 | Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1 | Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2 | Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet | Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1 | Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet
Started | 3 | 3 | 4 | 4 | 4 | 4
Completed | 3 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Methylprednisolone 32 mg Tablet, Formulation 1, Formulation 2 | Methylprednisolone 32 mg Tablet, Formulation 2, Formulation 1 | Methylprednisolone Formulation 1, 32 mg Tablet, Formulation 2 | Methylprednisolone Formulation 1, Formulation 2, 32 mg Tablet | Methylprednisolone Formulation 2, 32 mg Tablet, Formulation 1 | Methylprednisolone Formulation 2, Formulation 1, 32 mg Tablet
Started | 3 | 3 | 4 | 4 | 4 | 4
Completed | 3 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants randomized to receive methylprednisolone 32 mg tablet first, formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) first and formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 12, 16 and 24 hours (hrs) post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized participants who were treated and had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Methylprednisolone 32 mg Tablet: Single oral dose of methylprednisolone 32 mg tablet on Day 1 of any of the three intervention periods.
- Methylprednisolone 32 mg Micronized API: Single dose of formulation 1: methylprednisolone oral suspension 4 mg/mL at 32 mg (Micronized API) on Day 1 of any of the three intervention periods.
- Methylprednisolone 32 mg Sieve Cut API: Single dose of formulation 2: methylprednisolone oral suspension 4 mg/mL at 32 mg (Sieve cut API) on Day 1 of any of the three intervention periods.
Arm/Group | Methylprednisolone 32 mg Tablet | Methylprednisolone 32 mg Micronized API | Methylprednisolone 32 mg Sieve Cut API
Number analyzed (Participants) | 24 | 22 | 23
ng*hr/mL | 1286.00 (385.27) | 1204.00 (394.65) | 1180.00 (355.26)
Statistical Analysis 1: Comparison: Methylprednisolone 32 mg Tablet vs Methylprednisolone 32 mg Micronized API; Natural log transformed AUC (0 - ∞) of methylprednisolone was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 92.11, 90% CI 2-sided [88.23 to 96.15]
Statistical Analysis 2: Comparison: Methylprednisolone 32 mg Tablet vs Methylprednisolone 32 mg Sieve Cut API; Natural log transformed AUC (0 - ∞) of methylprednisolone was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 90.22, 90% CI 2-sided [86.49 to 94.11]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 12, 16 and 24 hrs post-dose
Population: PK parameter analysis population included all randomized participants who were treated and had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methylprednisolone 32 mg Tablet | Methylprednisolone 32 mg Micronized API | Methylprednisolone 32 mg Sieve Cut API
Number analyzed (Participants) | 24 | 22 | 23
ng/mL | 289.00 (60.42) | 279.10 (82.91) | 246.20 (66.05)
Statistical Analysis 1: Comparison: Methylprednisolone 32 mg Tablet vs Methylprednisolone 32 mg Micronized API; Natural log transformed Cmax of methylprednisolone was analyzed using mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of adjusted geometric means = 94.76, 90% CI 2-sided [88.06 to 101.98]
Statistical Analysis 2: Comparison: Methylprednisolone 32 mg Tablet vs Methylprednisolone 32 mg Sieve Cut API; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio of adjusted geometric means = 83.89, 90% CI 2-sided [78.06 to 90.17]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 12, 16 and 24 hrs post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Methylprednisolone 32 mg Tablet | Methylprednisolone 32 mg Micronized API | Methylprednisolone 32 mg Sieve Cut API
Number analyzed (Participants) | 24 | 22 | 23
hr | 2.00 [1.00 to 4.00] | 1.00 [0.50 to 4.00] | 2.00 [1.00 to 3.00]

4. Secondary Outcome: Plasma Decay Half-life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 12, 16 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Methylprednisolone 32 mg Tablet | Methylprednisolone 32 mg Micronized API | Methylprednisolone 32 mg Sieve Cut API
Number analyzed (Participants) | 24 | 22 | 23
hr | 2.43 (0.39) | 2.42 (0.37) | 2.45 (0.35)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Methylprednisolone 32 mg Tablet | Methylprednisolone 32 mg Micronized API | Methylprednisolone 32 mg Sieve Cut API
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 4/24 | 0/22 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylprednisolone 32 mg Tablet (N=24) | Methylprednisolone 32 mg Micronized API (N=22) | Methylprednisolone 32 mg Sieve Cut API (N=23)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.